CLINICAL TRIAL: NCT01082042
Title: Exercising With Computers in Later Life (EXCELL) - Pilot and Feasibility Study of the Nintendo® WiiFit in Community-dwelling Fallers
Brief Title: Exercising With Computers in Later Life
Acronym: EXCELL
Status: Completed | Type: Observational
Sponsor: NHS Grampian (Other Government)
Collaborators: British Geriatrics Society (Other)
Responsible Party: Dr Marie Williams, NHS Grampian
Other Study IDs: BGS05/2008
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2009-06

CONDITIONS: Accidental Falls; Exercise
Keywords: Balance, postural; Aged, over 70; Exercise; Accidental falls
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard Care: Individuals who attended the local falls group
- Intervention group: Individuals who undertook the 12 week exercise (Nintendo WiiFit) intervention

SUMMARY:
This is a pilot study to assess whether balance training with the Nintendo® Wii is comparable to a physiotherapist-led falls group in terms of improvement in balance. The acceptability of the Nintendo® Wii will also be assessed.

DETAILED DESCRIPTION:
The population is ageing and as a result medical staff and allied health professionals are likely to see an increase in the number of patients with falls. Community dwelling individuals over 65 fall at a rate of 30% per year. This risk increases with advancing age. Falls have significant consequences for both the individual and the population as a whole. Falls risk increases with age due to increased body sway, a reduction in reaction times, deterioration in the efficiency of the walking pattern and diminished balance.

People who fall should be referred for multidisciplinary falls assessment. Locally, patients are assessed by the multidisciplinary team and, if appropriate, attend falls group. This group consists of a 12 week exercise program to improve balance and muscle strength (patients attend the group up to 3 times weekly). Previously trials have shown variable compliance with exercise programs but locally compliance is felt to be good. Falls groups aim to reduce falls through the benefits of exercise; improvement in muscle strength,balance, general fitness and well being. It has been shown that exercise has statistically significant beneficial effects on balance.

Due to advances in technology, equipment has been produced to improve balance on both the medical and commercial market. There is a large variability in cost between this equipment with commercial prices being much lower. The Wii has been very successful in encouraging sedentary youths to partake in exercise (all be it in a limited form). WiiFit is a specifically designed "game" for the Wii to improve balance with an element of entertainment value.

This project is important due the large number of falls that occur in the community and the significant impact this has on an under resourced NHS. It is timely because the WiiFit has only just been introduced into the market. Through the use of a Wii, balance training may be more enjoyable and as a result elderly community dwellers may be more likely to participate in exercise programmes. The Wii is considerably cheaper than the medical alternatives and if an improvement can be shown in post-intervention balance assessments, then we have to consider whether the use of similar equipment should be instituted in falls groups.

ELIGIBILITY:
Inclusion Criteria:

* age 70 years or older
* living locally in the community (in either sheltered accommodation or own home
* fallen at least once in the preceding 12 months
* abbreviated mental test (AMT) of seven or over

Exclusion Criteria:

* wheelchair bound
* people living in a care home or long-term hospital care.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Standard Care: The standard care group was recruited from the local falls group that is run from the local Medicine for the Elderly Department.
  Intevention Group: Participants were recruited following a publicity campaign.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Improvement in formal balance score | 4 weeks and 12 weeks following the exercise intervention
  Berg and Tinetti balance scores

SECONDARY OUTCOMES:
Acceptability of the Nintendo WiiFit in community-dwelling older fallers | 12 weeks
  Individual interview and completion of the Attitudes to Falls-Related Interventions Scale (AFRIS)
Participants degree of concern about falling in certain situations following the intervention | 4 weeks and 12 weeks
  Falls Efficacy Scale - International (FES-I)

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Williams, MBChB, Principal Investigator — NHS Grampian
Locations (1):
- Department of Medicine for the Elderly, Woodend Hospital, Aberdeen, Aberdeenshire, United Kingdom

REFERENCES:
- [Derived] Williams MA, Soiza RL, Jenkinson AM, Stewart A. EXercising with Computers in Later Life (EXCELL) - pilot and feasibility study of the acceptability of the Nintendo(R) WiiFit in community-dwelling fallers. BMC Res Notes. 2010 Sep 13;3:238. doi: 10.1186/1756-0500-3-238. PMID 20831836